CLINICAL TRIAL: NCT06222944
Title: A Multi-Center, Multi-Cohort Study of the Efficacy and Safety of Anlotinib, TQB2450, and Albumin-bound Paclitaxel in CLDN18.2-regimen-failed Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Brief Title: Anlotinib, TQB2450 (PD-L1 Inhibitor), and Albumin-bound Paclitaxel Regimens in the Treatment of GC/GEJA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-GA001
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Adenocarcinoma of Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — anlotinib; Albumin-Bound Paclitaxel; Taxes; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib, TQB2450 and Albumin-bound Paclitaxel (Experimental): * Cohort 1: Anlotinib + albumin-bound paclitaxel;
  * Cohort 2: TQB2450 + albumin-bound paclitaxel;
  * Cohort 3: Anlotinib + TQB2450 + albumin-bound paclitaxel.
  Anlotinib: 12mg PO, QD, D1-14, Q3W;
  TQB2450: 1200 mg, IV, D1, Q3W;
  Albumin-bound paclitaxel: 125mg/m2 IV Day 1,8, Q3W.
  Until disease progression or intolerable toxicity or patient withdrawal of consent.
  Interventions: Drug: Anlotinib; Drug: TQB2450; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: Anlotinib — Anlotinib: 12mg PO, QD, D1-14, Q3W;
  Other Names: Anlotinib Hydrochloride Capsule
Drug: TQB2450 — TQB2450: 1200 mg, IV, D1, Q3W
Drug: Albumin-Bound Paclitaxel — 125mg/m2 IV D1,8，Q3W
  Other Names: Paclitaxel (albumin-bound); Paclitaxel for injection(Albumin Bound)

SUMMARY:
This study aims to assess the efficacy and safety of a combination therapy consisting of Anlotinib, TQB2450 (a PD-L1 inhibitor), and Albumin-bound Paclitaxel regimens in patients with advanced gastric cancer (GC) or gastroesophageal junction adenocarcinoma (GEJA) who have failed the previous treatment with Claudin18.2 (CLDN18.2)-related regimens.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily join this study, sign the informed consent form, and have good compliance;
* Pathologically (histologically or cytologically) confirmed HER2/neu-negative (or HER2/neu status unclear) advanced gastric cancer or gastroesophageal junction adenocarcinoma;
* Patients who have failed first-line treatment with CLDN18.2-related regimen (CLDN18.2 drugs include CLDN18.2 monotherapy, CLDN18.2 dual therapy, CLDN18.2 ADC or CLDN18.2 CART therapy, treatment regimen includes CLDN18.2 combined with chemotherapy or immunotherapy or other systemic therapy) and the time from the end of the last treatment with CLDN18.2-related drugs is more than two weeks;
* According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, at least one measurable lesion, which can be accurately measured in at least one direction (the maximum diameter needs to be recorded) by magnetic resonance imaging (MRI) or computed tomography (CT), with the longest diameter at baseline ≥10 mm (if it is a lymph node, the short diameter is required to be ≥15 mm); the measurable lesions should not have received local treatment such as radiotherapy (lesions in the previous radiotherapy area, if confirmed to have progressed and meet the RECIST 1.1 criteria, can also be selected as target lesions);
* Male or female patients aged ≥18 years and ≤75 years;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0-1;
* Expected survival ≥3 months;
* Adequate organ function, requiring the following laboratory test values at screening:

  * Hemoglobin (HB) ≥80g/L (no blood transfusion within 14 days);
  * Absolute neutrophil count (ANC) ≥1.5×109/L;
  * Platelet count (PLT) ≥75×109/L (no use of interleukin 11 or TPO within 14 days);
  * White blood cell count (WBC) ≥3.0×109/L (no use of granulocyte stimulating factor within 14 days).
  * Serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN);
  * ALT and AST ≤2.5 ULN, if there is liver metastasis, then ALT and AST ≤5×ULN;
  * Creatinine (Cr) ≤1.5 ULN or creatinine clearance rate (CCr) ≥60ml/min, (Cockcroft-Gault formula);
  * Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  * Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%);
  * Cardiac enzyme spectrum: within normal range;
* Women of childbearing age must take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and must be non-lactating patients. Serum or urine pregnancy test negative within 7 days before enrollment in the study, or meet one of the following criteria to prove that there is no risk of pregnancy:

  * a) Postmenopausal is defined as age over 50 years and amenorrhea for at least 12 months after stopping all exogenous hormone replacement therapy;
  * b) Women under 50 years of age, if amenorrhea for 12 months or more after stopping all exogenous hormone therapy, and luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the laboratory postmenopausal reference range, can also be considered as postmenopausal;
  * c) Have undergone irreversible sterilization surgery, including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but excluding bilateral tubal ligation; For men, they must agree to use appropriate methods of contraception or have undergone surgical sterilization during the trial and 8 weeks after the last administration of the trial drug;

Exclusion Criteria:

* For cohort 1, patients who have previously received anlotinib hydrochloride treatment or other anti-angiogenic small molecule tyrosine kinase inhibitors (TKIs) within 6 months. Patients who have stopped treatment with other anti-angiogenic small molecule TKIs for more than 6 months are allowed to enroll; For cohort 2 and cohort 3, patients who have received PD-L1 immune checkpoint inhibitor treatment in the first line are excluded, but patients who have received PD-1 or CTLA-4 immune checkpoint inhibitor treatment in the first line are allowed, if they have any of the following immune-related medical history and treatment history, they are excluded:

  * Have any active autoimmune disease or history of autoimmune disease (such as but not limited to autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; requiring bronchodilators for medical intervention of asthma); but the following patients are allowed to enroll: vitiligo, psoriasis, alopecia that do not require systemic treatment, type I diabetes that is well controlled, hypothyroidism that has normal thyroid function after replacement therapy;
  * Diagnosed with immunodeficiency or receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy (dose >10mg/day of prednisone or other equivalent hormones), and continuing to use it within 2 weeks before the first administration;
  * Received any live vaccine, attenuated vaccine (including anti-infective vaccines, such as influenza vaccine, varicella vaccine, etc.), or inactivated vaccine within 4 weeks before enrollment and plan to receive live vaccine/attenuated vaccine/inactivated vaccine during the study; used systemic immunostimulants (including but not limited to interferon and IL-2) within 2 weeks before the start of the study treatment;

For Cohort 3, patients who have previously received anlotinib hydrochloride or other anti-angiogenic small molecule tyrosine kinase inhibitors (TKIs) within 6 months. Patients who have stopped treatment with other anti-angiogenic small molecule TKIs for more than 6 months are allowed to enroll;

* Patients who have received anti-tumor treatment with traditional Chinese medicine within the past two weeks (the traditional Chinese medicine contains the following medicinal materials such as Brucea javanica, Coix seed, Lentinan, Cantharidin, Toad skin, Astragalus, Sophora, Ugonin, Chebula, Icariin, etc.), but patients who have stopped taking anti-tumor treatment with traditional Chinese medicine for more than two weeks are allowed to enroll;
* Patients who have received ≥1 other systemic systemic anti-tumor treatment (including but not limited to chemotherapy, immunotherapy, targeted therapy, and other systemic treatment regimens) after failing CLDN18.2-related regimen treatment, but palliative local treatment (including radiotherapy and other local treatment regimens) for local lesions (non-target lesions) >two weeks later are allowed to enroll;
* Patients who have previously received allogeneic bone marrow transplantation or organ transplantation;
* Congenital pulmonary fibrosis, drug-induced pneumonia, organizing pneumonia, or CT-confirmed active pneumonia;
* Patients with symptomatic central nervous system metastases and/or carcinomatous meningitis. Patients with a history of central nervous system metastases or spinal cord compression, if they have received treatment and stopped using anticonvulsants and steroids 4 weeks before the first administration of the study and have clinically stable performance, can enroll in the study;
* ≥ NCI CTCAE grade 2 peripheral neuropathy;
* Infection requiring antibiotics within 14 days before the start of the trial;
* Patients with bone metastases at risk of paraplegia;
* Patients with any severe and/uncontrolled disease, including:

  * Patients with poor blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg); patients with grade II or higher myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥480ms); patients with III-IV heart failure according to NYHA criteria or cardiac ultrasound examination suggesting left ventricular ejection fraction (LVEF) <50%;
  * Poorly controlled diabetes (fasting blood glucose (FBG) >10mmol/L);
  * Urinalysis suggests urine protein ≥++, and 24-hour urine protein quantification >1.0 g is confirmed;
* Received major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks before the study, or expected to need major surgery during the study treatment, or non-diagnostic surgery within 4 weeks before the start of the trial;
* History of gastrointestinal perforation and/or fistula within 6 months before enrollment; or history of arterial/venous thromboembolic events, such as cerebrovascular accident (stable cerebral infarction excluded by researcher evaluation), deep vein thrombosis, and pulmonary embolism;
* Clinically significant pleural effusion, including any pleural effusion that can be found by physical examination, pleural effusion that has been treated in the past or still needs treatment. Patients with only a small amount of pleural effusion shown by imaging but no symptoms, and who do not need treatment according to the researcher's evaluation, can be enrolled;
* Body mass index (BMI) <17.0 kg/m² or weight loss of ≥10% within 2 months before screening;
* Patients with a history of psychotropic drug abuse and unable to quit or have mental disorders;
* Patients with active hepatitis B or hepatitis C, HIV-positive patients, patients with active tuberculosis;
* CT suggests definite ulcerative lesions, or occult blood in stool ++ or above;
* History of abnormal bleeding (except epistaxis) within 1 month before enrollment;
* History of other primary malignant tumors, except for the following: 1) Malignant tumors that have been completely remitted for at least 2 years before enrollment and do not require other treatment during the study; 2) Non-melanoma skin cancer or malignant melanocytic nevus that have been adequately treated and have no evidence of disease recurrence; 3) In situ carcinoma that has been adequately treated and has no evidence of disease recurrence;
* Pregnant or lactating female patients;
* According to the researcher's judgment, patients with severe accompanying diseases that endanger the patient's safety or affect the patient's completion of the study;
* Participated in other trials within 30 days before the start of the trial, or plan to participate in other trials during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
ORR | Baseline to CR/PR, about 12 months
  Objective Response Rate (ORR) is defined as the percentage of participants who achieve either a complete response (CR) or a partial response (PR) according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
DCR | Baseline to CR/PR, about 16 months
  Disease Control Rate (DCR) is defined as the percentage of participants with complete response (CR), partial response (PR), or stable disease (SD).
PFS | Baseline to CR/PR, about 16 months
  Progression-free survival (PFS) is the time elapsed between treatment initiation and tumor progression or death from any cause based on the RECIST 1.1 criteria.
OS | Baseline to CR/PR, about 20 months
  Overall Survival (OS) is defined as the time from the first dose of study drugs to the time of death from any cause.
Adverse events | Baseline to CR/PR, about 20 months
  The adverse events (AEs) were assessed by investigators according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China